CLINICAL TRIAL: NCT00401635
Title: Phase II Multicentered Study of First-Line Chemotherapy for Advanced or Recurrent Endometrial Carcinoma With the Combination of Carboplatin and Liposomal Doxorubicin
Brief Title: END-1: First Line Chemotherapy for Advanced or Recurrent Endometrial Carcinoma With Carboplatin and Liposomal Doxorubicin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: END-1
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-09

CONDITIONS: Endometrial Cancer
Keywords: advanced; recurrent; chemotherapy; first-line
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — liposomal doxorubicin; Carboplatin

INTERVENTIONS:
Drug: liposomal doxorubicin
Drug: carboplatin

SUMMARY:
The purpose of this study is to evaluate activity and toxicity of the combination of carboplatin and liposomal doxorubicin as first-line chemotherapy of patients with advanced or recurrent endometrial carcinoma.

DETAILED DESCRIPTION:
Treatment is planned with carboplatin AUC 5 given IV on day 1 and liposomal doxorubicin 40 mg/m2 given IV on day 1, with treatment repeated every 28 days. Delays in treatment administration and dose reductions have been planned according to toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic / histologic diagnosis of endometrial carcinoma
* Indication for chemotherapy
* Age 75 years or less
* Life expectancy of at least 3 months
* Measurable disease > 1 cm

Exclusion Criteria:

* Previous or concomitant malignant neoplasia (not including basocellular or spinocellular skin carcinoma or in-situ carcinoma of the uterine cervix, provided they are being adequately treated)
* Performance status (ECOG) > 2
* Previous chemotherapy treatment
* Heart disease (heart failure, myocardial heart attack within 6 months prior to randomization, atrioventricular block of any degree, serious arrhythmia)
* Leukocytes < 4000/mm3, platelets < 100000/mm3
* Impaired renal function (creatinine > o = 1.25 times the upper normal limit) or liver function (SGOT or SGPT > o = 1.25 times the upper normal limit)
* Present or suspected hemorrhagic syndromes
* Uncooperative and/or unreliable patients
* Patient's inability to access the center
* Refusal of informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2002-11

PRIMARY OUTCOMES:
Objective response rate (complete and partial responses)
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples
Locations (4):
- Italy (4):
  - Ospedale Fatebenefratelli, U.O. di Oncologia, Benevento, BN
  - Ospedale Pierantoni, Divisione di Oncologia Medica, Forlì, FO
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma, Roma
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli

REFERENCES:
- [Result] Pignata S, Scambia G, Pisano C, Breda E, Di Maio M, Greggi S, Ferrandina G, Lorusso D, Zagonel V, Febbraro A, Riva N, De Rosa V, Gallo C, Perrone F; Multicentre Italian Trials in Ovarian Cancer and Gynecologic Malignancies Group. A multicentre phase II study of carboplatin plus pegylated liposomal doxorubicin as first-line chemotherapy for patients with advanced or recurrent endometrial carcinoma: the END-1 study of the MITO (Multicentre Italian Trials in Ovarian Cancer and Gynecologic Malignancies) group. Br J Cancer. 2007 Jun 4;96(11):1639-43. doi: 10.1038/sj.bjc.6603787. Epub 2007 May 8. PMID 17486128